CLINICAL TRIAL: NCT02111915
Title: Thinking Healthy Program - Peer Delivered in Pakistan
Brief Title: Thinking Healthy Program - Peer Delivered (Pakistan)
Acronym: THPP-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Principal Investigator, Atif Rahman, Prof Atif Rahman, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: THPP-P MH095687; 1U19MH095687-01 (NIH)
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Unipolar Depression
Keywords: Maternal depression
MeSH Terms: conditions — Depressive Disorder | interventions — meso-tetra-(4-hydroxyphenyl)porphyrin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (EUC) (Other): EUC will comprise communicating the results to the mother's Lady Health Worker and medical officer (MO) at the Basic Health Unit (BHU) of her area, providing the MO with the WHO mental health gap (mhGAP) guidelines for the treatment of depression, and providing guidance on referral of depressed mothers to mental health services
  Interventions: Other: EUC
- THPP-P (Experimental): Trial participant s who are in the THPP group will receive, in addition to EUC, 14 sessions of THPP (simplified cognitive behaviour therapy) starting from their recruitment in the third trimester until up to 5 months after child birth.
  Interventions: Behavioral: THPP-P; Other: EUC

INTERVENTIONS:
Behavioral: THPP-P — Trial participant s who are in the THPP group will receive, in addition to Enhanced Usual Care (EUC), 14 sessions of THPP (simplified cognitive behaviour therapy) starting from their recruitment in the third trimester until up to 5 months after child birth.
  Other Names: Thinking Healthy Program : Peer Delivered - Pakistan
  Arms: THPP-P
Other: EUC — EUC will comprise communicating the results to the mother's Lady Health Worker and medical officer (MO) at the Basic Health Unit (BHU) of her area, providing the MO with the WHO mental health gap (mhGAP) guidelines for the treatment of depression, and providing guidance on referral of depressed mothers to mental health services.
  Other Names: Enhanced Usual Care

SUMMARY:
The rates of perinatal depression in South Asian women are reported to be amongst the highest in the world, ranging from 18%-30% in urban areas and 28%-36% in rural areas. In addition to its profound impact on women's health, disability and functioning, perinatal depression is associated with poor child health outcomes such as pre-term birth, infant under-nutrition and stunting. There is robust evidence that perinatal depression can be effectively managed with psychological treatments delivered by non-specialist health care workers. Our previous research conducted in Pakistan led to the development of the Thinking Healthy Program (THP). THP is a psychological treatment delivered by community health workers (CHWs) which more than halved the rate of perinatal depression among mothers and led to significant improvements in child health outcomes. To enhance access to such evidence-based psychological treatments, there is a need to examine the potential role of other human resources such as lay persons in delivering psychological treatments such as THP in poor resource settings.

DETAILED DESCRIPTION:
Objectives To evaluate the effectiveness and cost-effectiveness of THP delivered by peers (the Thinking Healthy Program - Peer delivered in Rawalpindi, Pakistan; THPP-P) over the duration of 6 months. Peers will be healthy mothers who live in the same community as potential trial participants (TPs).

Study design and outcomes Single-blind stratified cluster randomized controlled trial in Rawalpindi, Pakistan (rural area) involving 40 clusters (560 women). TPs will not be blinded to treatment allocation. TPs include all pregnant women in their third trimester of pregnancy who are identified through the list of their local community health worker (Lady Health Worker or LHW). Those who are eligible will be invited to participate in screening for depression; mothers who consent will be screened for depression with a locally validated version of the Patient Health Questionnaire (PHQ-9). TPs who screen positive (PHQ-9 score ≥ 10) receive enhanced usual care (EUC) or THPP+EUC. The primary outcome measures will be remission (i.e. recovery from depression) and reduction in depressive symptoms, both assessed by the PHQ-9 at 6 months post child birth. Secondary outcomes are depressive symptoms and remission at 3 months (PHQ-9), maternal disability at 3 and 6 months post child birth (measured with the WHO-DAS), improved maternal support (measured with MSPSS) at 3 and 6 months post child birth, breastfeeding rates and infant weight and height of children at 3 and 6 months. Outcomes will be analysed on an intention to treat basis.

Interventions EUC will comprise communicating the results to the mother's LHW and medical officer (MO) at the Basic Health Unit (BHU) of her area, providing the MO with the WHO mhGAP guidelines for the treatment of depression, and providing guidance on referral of depressed mothers to mental health services. TPs who are in the THPP group will receive, in addition, 14 sessions of THPP starting from their recruitment in the third trimester until up to 5 months after child birth. Sessions will be delivered by peers on an individual and group basis at a location of convenience to the TPs (usually at their own homes).

Implications THPP has the potential to advance knowledge of the extent to which task-shifting of the delivery of evidence-based psychological treatments can be extended to peers in the community. If effectiveness is observed, this approach offers a potential opportunity to access a vast untapped human resource for maternal mental health care and addresses a major barrier in global mental health - the lack of skilled and motivated human resources in the formal health sector - offering a new avenue for the scaling up of evidence-based psychological treatments in low resourced settings.

ELIGIBILITY:
Inclusion Criteria:

* Depressive disorder (PHQ-9 (>10 score)),
* In the 3rd trimester of pregnancy,
* Aged 18 years and over,
* Intending to reside in the study area for the entire duration of the study.

Exclusion criteria:

* Mothers requiring immediate inpatient care for any reason (medical or psychiatric),
* Mothers who do not speak any of the following languages: Urdu, Punjabi, Potohari or English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Remission (i.e. recovery from depression) | 6 months post child birth
  Measured with the Patient Health Questionnaire- 9 (PHQ-9)

SECONDARY OUTCOMES:
Remission (i.e. recovery from depression) | 3 months post child birth
  Measured with the Patient Health Questionnaire-9 (PHQ-9)
Maternal disability | 3 and 6 months post child birth
  Measured with the World Health Organization's Disability Assessment Schedule (WHO-DAS)
Maternal support | 3 and 6 months post child birth
  Measured with the Multidimensional Scale of Perceived Social Support (MSPSS)
Breastfeeding rates | 3 and 6 months post child birth
Infant height | 3 and 6 months post child birth

CONTACTS AND LOCATIONS:
Overall Officials: Atif Rahman, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Human Development Research Foundation, Islamabad, Pakistan

REFERENCES:
- [Derived] LeMasters K, Bates LM, Chung EO, Gallis JA, Hagaman A, Scherer E, Sikander S, Staley BS, Zalla LC, Zivich PN, Maselko J. Adverse childhood experiences and depression among women in rural Pakistan. BMC Public Health. 2021 Feb 25;21(1):400. doi: 10.1186/s12889-021-10409-4. PMID 33632175
- [Derived] Vanobberghen F, Weiss HA, Fuhr DC, Sikander S, Afonso E, Ahmad I, Atif N, Bibi A, Bibi T, Bilal S, De Sa A, D'Souza E, Joshi A, Korgaonkar P, Krishna R, Lazarus A, Liaqat R, Sharif M, Weobong B, Zaidi A, Zuliqar S, Patel V, Rahman A. Effectiveness of the Thinking Healthy Programme for perinatal depression delivered through peers: Pooled analysis of two randomized controlled trials in India and Pakistan. J Affect Disord. 2020 Mar 15;265:660-668. doi: 10.1016/j.jad.2019.11.110. Epub 2019 Nov 23. PMID 32090783
- [Derived] LeMasters K, Andrabi N, Zalla L, Hagaman A, Chung EO, Gallis JA, Turner EL, Bhalotra S, Sikander S, Maselko J. Maternal depression in rural Pakistan: the protective associations with cultural postpartum practices. BMC Public Health. 2020 Jan 15;20(1):68. doi: 10.1186/s12889-020-8176-0. PMID 31941468
- [Derived] Scherer E, Hagaman A, Chung E, Rahman A, O'Donnell K, Maselko J. The relationship between responsive caregiving and child outcomes: evidence from direct observations of mother-child dyads in Pakistan. BMC Public Health. 2019 Feb 28;19(1):252. doi: 10.1186/s12889-019-6571-1. PMID 30819173
- [Derived] Sikander S, Ahmad I, Atif N, Zaidi A, Vanobberghen F, Weiss HA, Nisar A, Tabana H, Ain QU, Bibi A, Bilal S, Bibi T, Liaqat R, Sharif M, Zulfiqar S, Fuhr DC, Price LN, Patel V, Rahman A. Delivering the Thinking Healthy Programme for perinatal depression through volunteer peers: a cluster randomised controlled trial in Pakistan. Lancet Psychiatry. 2019 Feb;6(2):128-139. doi: 10.1016/S2215-0366(18)30467-X. PMID 30686386
- [Derived] Atif N, Krishna RN, Sikander S, Lazarus A, Nisar A, Ahmad I, Raman R, Fuhr DC, Patel V, Rahman A. Mother-to-mother therapy in India and Pakistan: adaptation and feasibility evaluation of the peer-delivered Thinking Healthy Programme. BMC Psychiatry. 2017 Feb 23;17(1):79. doi: 10.1186/s12888-017-1244-z. PMID 28231791
- [Derived] Turner EL, Sikander S, Bangash O, Zaidi A, Bates L, Gallis J, Ganga N, O'Donnell K, Rahman A, Maselko J. The effectiveness of the peer delivered Thinking Healthy Plus (THPP+) Programme for maternal depression and child socio-emotional development in Pakistan: study protocol for a three-year cluster randomized controlled trial. Trials. 2016 Sep 8;17(1):442. doi: 10.1186/s13063-016-1530-y. PMID 27608926
- [Derived] Sikander S, Lazarus A, Bangash O, Fuhr DC, Weobong B, Krishna RN, Ahmad I, Weiss HA, Price L, Rahman A, Patel V. The effectiveness and cost-effectiveness of the peer-delivered Thinking Healthy Programme for perinatal depression in Pakistan and India: the SHARE study protocol for randomised controlled trials. Trials. 2015 Nov 25;16:534. doi: 10.1186/s13063-015-1063-9. PMID 26604001